CLINICAL TRIAL: NCT01585766
Title: A Phase 1 Randomized Study of MEDI-551 in Subjects With Relapsing Forms of Multiple Sclerosis
Brief Title: Safety and Tolerability Study of MEDI-551, a B-cell Depleting Agent, to Treat Relapsing Forms of Multiple Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CD-IA-MEDI-551-1102
Record Dates: First submitted 2012-04-09; First posted 2012-04-26 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-02

CONDITIONS: Multiple Sclerosis, Relapsing Forms
Keywords: MAb, B cell, depletion, RMS
MeSH Terms: conditions — Multiple Sclerosis; Mycobacterium Infections, Nontuberculous | interventions — inebilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- MEDI-551 30 MG-IV (Experimental): Participants received a fixed IV dose of 30 milligram (mg) MEDI-551 infused on Days 1 and 15.
  Interventions: Drug: MEDI-551 30 MG-IV
- MEDI-551 60 MG-SC (Experimental): Participants received SC injection of 60 mg MEDI-551 on Day 1.
  Interventions: Drug: MEDI-551 60 MG-SC
- MEDI-551 100 MG-IV (Experimental): Participants received a fixed IV dose of 100 mg MEDI-551 infused on Days 1 and 15.
  Interventions: Drug: MEDI-551 100 MG-IV
- MEDI-551 300 MG-SC (Experimental): Participants received SC injection of 300 mg MEDI-551 on Day 1.
  Interventions: Drug: MEDI-551 300 MG-SC
- MEDI-551 600 MG-IV (Experimental): Participants received a fixed IV dose of 600 mg MEDI-551 infused on Days 1 and 15.
  Interventions: Drug: MEDI-551 600 MG-IV
- PLACEBO-IV-SC (Placebo Comparator): Participants received either a fixed IV dose of placebo matching with MEDI- 551 on Days 1 and 15 or SC injection on Day 1.
  Interventions: Drug: PLACEBO-IV-SC

INTERVENTIONS:
Drug: MEDI-551 30 MG-IV — Participants received a fixed IV dose of 30 milligram (mg) MEDI-551 infused on Days 1 and 15.
  Arms: MEDI-551 30 MG-IV
Drug: MEDI-551 60 MG-SC — Participants received SC injection of 60 mg MEDI-551 on Day 1.
  Arms: MEDI-551 60 MG-SC
Drug: PLACEBO-IV-SC — Participants received either a fixed IV dose of placebo matching with MEDI- 551 on Days 1 and 15 or SC injection on Day 1
  Arms: PLACEBO-IV-SC
Drug: MEDI-551 100 MG-IV — Participants received a fixed IV dose of 100 mg MEDI-551 infused on Days 1 and 15.
  Arms: MEDI-551 100 MG-IV
Drug: MEDI-551 300 MG-SC — Participants received SC injection of 300 mg MEDI-551 on Day 1.
  Arms: MEDI-551 300 MG-SC
Drug: MEDI-551 600 MG-IV — Participants received a fixed IV dose of 600 mg MEDI-551 infused on Days 1 and 15.
  Arms: MEDI-551 600 MG-IV

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of ascending intravenous (IV) and subcutaneous (SC) doses of MEDI-551 in adult subjects with relapsing forms of multiple sclerosis (MS).

DETAILED DESCRIPTION:
This is a Phase 1, multicenter, multinational, randomized, blinded, placebo-controlled, dose-escalation study to evaluate the safety and tolerability of IV and SC doses of MEDI-551 in adult subjects with relapsing forms of MS.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed relapsing form of MS (ie, RRMS, SPMS, PRMS, or CIS) according to revised 2010 McDonald criteria and MRI brain lesions consistent with MS on screening
* At least 1 documented relapse within the past 3 years prior to screening
* EDSS between 0.0 and 6.5 at screening
* Have no more than 20 Gd-enhancing T1 brain lesions detected by cranial MRI scan

Exclusion Criteria:

* Subjects with impaired renal function
* Major surgery within 8 weeks of the screening visit
* Subjects who are unable to undergo cranial MRI scan
* A history of hypersensitivity to Gd-containing MRI contrast agents
* Has received within 1 year prior to screening: monoclonal antibodies, experimental B-cell depleting agents, or treatment with natalizumab (Tysabri) for greater than 3 months
* Receiving monthly methylprednisone or equivalent glucocorticoid for disease modification of a relapsing form of MS
* Known sensitivity to acetaminophen/paracetamol, diphenhydramine or equivalent antihistamine, methylprednisolone or equivalent glucocorticoid, or to any component of the investigational drug
* Diagnosis of PPMS, neuromyelitis optica, or other non-MS variant of neuro-inflammatory or demyelinating diseases
* Any history of opportunistic infection or the presence of active infection within two months prior to screening or any herpes zoster infection that has not resolved within 12 weeks prior to screening
* Any clinically significant findings during the screening phase, including physical, neurological, laboratory, or ECG examination as per protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-04-24 (Actual); Primary Completion 2015-01-02 (Actual); Study Completion 2016-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Armando Flor, Study Director — MedImmune LLC
Locations (16):
- United States (9):
  - Research Site, Scottsdale, Arizona
  - Research Site, Long Beach, California
  - Research Site, Sacramento, California
  - Research Site, Denver, Colorado
  - Research Site, Tampa, Florida
  - Research Site, Marlton, New Jersey
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cordova, Tennessee
  - Research Site, Houston, Texas
- Poland (2):
  - Research Site, Katowice
  - Research Site, Szczecin
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Girona
  - Research Site, Seville
- Ukraine (2):
  - Research Site, Donetsk
  - Research Site, Kyiv

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 30 Jul 2012 to 20 Jun 2016 in United States, Poland, Spain, and Ukraine.
Pre-assignment Details: A total of 56 participants were screened in this study. Out of which 28 participants were enrolled and randomized into the study.
Groups:
- PLACEBO-IV-SC: Participants received either a fixed IV dose of placebo matching MEDI-551 on Days 1 and 15 or SC injection on Day 1.
Period: Overall Study
Arm/Group | PLACEBO-IV-SC | MEDI-551 30 Mg-IV | MEDI-551 60 Mg-SC | MEDI-551 100 Mg-IV | MEDI-551 300 Mg-SC | MEDI-551 600 Mg-IV
Started | 7 | 5 | 3 | 4 | 3 | 6
Completed | 7 | 3 | 1 | 4 | 3 | 6
Not Completed | 0 | 2 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population is defined as all participants who received any amount of study drug. One participant in the 30 mg IV dose cohort received an incorrect dose of study drug due to kits not administered according to the IVRS; the participant received MEDI-551 100 mg IV instead of 30 mg on Day 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | PLACEBO-IV-SC | MEDI-551 30 Mg-IV | MEDI-551 60 Mg-SC | MEDI-551 100 Mg-IV | MEDI-551 300 Mg-SC | MEDI-551 600 Mg-IV | Total
Number analyzed (Participants) | 7 | 5 | 3 | 4 | 3 | 6 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.0 (15.9) | 42.4 (7.8) | 46.7 (16.3) | 46.5 (13.8) | 56.0 (6.1) | 44.2 (10.1) | 45.4 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 2 | 3 | 2 | 3 | 19
  Male | 1 | 2 | 1 | 1 | 1 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A TEAE were the events between administration of study drug (Day 1) and Day 169 that were absent before treatment or that worsened relative to pre-treatment state. The AEs were summarized using Medical Dictionary for Regulatory Activities version 19.0
Time Frame: From study drug administration (Day 1) through the end of treatment period (Day 169)
Population: Safety Population is defined as all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | PLACEBO-IV-SC | MEDI-551 30 Mg-IV | MEDI-551 60 Mg-SC | MEDI-551 100 Mg-IV | MEDI-551 300 Mg-SC | MEDI-551 600 Mg-IV
Number analyzed (Participants) | 7 | 5 | 3 | 4 | 3 | 6
Participants | 6 | 5 | 3 | 3 | 3 | 6

2. Primary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (TESAEs)
Description: A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death, life-threatening, initial or prolonged inpatient hospitalization, persistent or significant disability or incapacity, congenital anomaly or birth defect in the offspring of a participant who received the study drug. The TESAEs were the events between administration of study drug (Day 1) and long term follow up period (up to 18 months after early discontinuation visit or 24-week treatment period) that were absent before treatment or that worsened relative to pre-treatment state. The AEs were summarized using Medical Dictionary for Regulatory Activities version 19.0
Time Frame: From study drug administration (Day 1) through the long term follow up period (up to 18 months after early discontinuation visit or 24 week treatment period).
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | PLACEBO-IV-SC | MEDI-551 30 Mg-IV | MEDI-551 60 Mg-SC | MEDI-551 100 Mg-IV | MEDI-551 300 Mg-SC | MEDI-551 600 Mg-IV
Number analyzed (Participants) | 7 | 5 | 3 | 4 | 3 | 6
Participants | 1 | 1 | 0 | 0 | 1 | 1

3. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities Reported as TEAEs
Description: Any clinically significant change in laboratory evaluations were recorded as AEs. The following parameters were analyzed for laboratory evaluations: haematology, serum chemistry, and urinalysis. Number of participants with TEAEs related to laboratory evaluations were reported.
Time Frame: From study drug administration (Day 1) through the end of treatment period (Day 169)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | PLACEBO-IV-SC | MEDI-551 30 Mg-IV | MEDI-551 60 Mg-SC | MEDI-551 100 Mg-IV | MEDI-551 300 Mg-SC | MEDI-551 600 Mg-IV
Number analyzed (Participants) | 7 | 5 | 3 | 4 | 3 | 6
Participants
  Hematology- Anaemia | 1 | 0 | 0 | 0 | 0 | 0
  Hematology- White blood cell count decreased | 0 | 0 | 0 | 1 | 0 | 0
  Serum chemistry- Liver function test increased | 0 | 1 | 0 | 0 | 0 | 0
  Serum chemistry- Hyponatraemia | 0 | 0 | 0 | 0 | 0 | 1

4. Primary Outcome: Number of Participants With Vital Sign Abnormalities Reported as TEAEs
Description: Vital sign parameters included blood pressure, temperature, pulse rate, and respiratory rate. The number of participants with TEAEs related to vital signs in participants were reported.
Time Frame: From study drug administration (Day 1) through the end of treatment period (Day 169)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | PLACEBO-IV-SC | MEDI-551 30 Mg-IV | MEDI-551 60 Mg-SC | MEDI-551 100 Mg-IV | MEDI-551 300 Mg-SC | MEDI-551 600 Mg-IV
Number analyzed (Participants) | 7 | 5 | 3 | 4 | 3 | 6
Participants
  Blood pressure increased | 1 | 0 | 1 | 0 | 0 | 2
  Blood pressure decreased | 0 | 0 | 1 | 0 | 0 | 0
  Tachycardia | 0 | 0 | 1 | 0 | 0 | 0

5. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) of MEDI-551
Description: The time to reach the maximum observed serum concentration of MEDI-551.
Time Frame: Predose (Day 1) and Postdose (IV Cohorts only), Days 4 (SC Cohorts only), 8, 15 Predose and Postdose (IV Cohorts only), 29, 57, 85, 113, 141, and 169
Population: Safety Population
Measure: Median (Full Range); unit: Day
Arm/Group | MEDI-551 30 Mg-IV | MEDI-551 60 Mg-SC | MEDI-551 100 Mg-IV | MEDI-551 300 Mg-SC | MEDI-551 600 Mg-IV
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 6
Day | 0.14 [0.11 to 0.19] | 2.98 [2.87 to 6.97] | 0.07 [0.01 to 0.11] | 7.92 [7.82 to 8.02] | 0.12 [0.11 to 0.18]

6. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of MEDI-551
Description: The maximum observed serum concentration (Cmax) of MEDI-551.
Time Frame: as for outcome 5
Population: Safety Population
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | MEDI-551 30 Mg-IV | MEDI-551 60 Mg-SC | MEDI-551 100 Mg-IV | MEDI-551 300 Mg-SC | MEDI-551 600 Mg-IV
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 6
microgram per milliliter (mcg/mL) | 17.9 (13.2) | 6.67 (2.88) | 43.1 (11.4) | 24.7 (9.37) | 248 (66.8)

7. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC 0-last) of MEDI-551
Description: The area under the concentration time curve from time 0 (dosing time) to the last measurable concentration (AUC 0-last) of MEDI-551.
Time Frame: as for outcome 5
Population: Safety Population
Measure: Mean (Standard Deviation); unit: microgram*day per milliliter(mcg*day/mL)
Arm/Group | MEDI-551 30 Mg-IV | MEDI-551 60 Mg-SC | MEDI-551 100 Mg-IV | MEDI-551 300 Mg-SC | MEDI-551 600 Mg-IV
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 6
microgram*day per milliliter(mcg*day/mL) | 436 (NA) — Standard deviation was not calculated due to limited sample size (n=2). Two out of five participants received only one dose and 1 participant had insufficient data. | 197 (92.6) | 1140 (278) | 788 (455) | 6850 (1340)

8. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Zero to Infinity (AUC 0-infinity) of MEDI-551
Description: The area under the concentration-time curve from dosing extrapolated to infinity (AUC 0-infinity) of MEDI-551.
Time Frame: as for outcome 5
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mcg*day/mL
Arm/Group | MEDI-551 30 Mg-IV | MEDI-551 60 Mg-SC | MEDI-551 100 Mg-IV | MEDI-551 300 Mg-SC | MEDI-551 600 Mg-IV
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 6
mcg*day/mL | 440 (NA) — Standard deviation was not calculated due to limited sample size (n=2). Two out of five participants received only one dose and 1 participant had insufficient data. | 201 (91.5) | 1150 (286) | 794 (453) | 6950 (1430)

9. Secondary Outcome: Dose Normalized Area Under the Plasma Concentration-time Curve From Zero to Infinity (AUC 0-infinity/D) of MEDI-551
Description: The AUC (0-infinity)/D is the area under concentration-time curve extrapolated to infinity post dose normalized by MEDI-551.
Time Frame: as for outcome 5
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mcg*day/mL/mg
Arm/Group | MEDI-551 30 Mg-IV | MEDI-551 60 Mg-SC | MEDI-551 100 Mg-IV | MEDI-551 300 Mg-SC | MEDI-551 600 Mg-IV
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 6
mcg*day/mL/mg | 7.34 (NA) — Standard deviation was not calculated due to limited sample size (n=2). Two out of five participants received only one dose and 1 participant had insufficient data. | 3.35 (1.52) | 5.75 (1.43) | 2.65 (1.51) | 5.79 (1.19)

10. Secondary Outcome: Clearance of MEDI-551
Description: Systemic clearance (CL) for MEDI-551 IV cohorts and apparent clearance (CL/F) for MEDI-551 SC cohorts were calculated
Time Frame: as for outcome 5
Population: Safety Population
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | MEDI-551 30 Mg-IV | MEDI-551 60 Mg-SC | MEDI-551 100 Mg-IV | MEDI-551 300 Mg-SC | MEDI-551 600 Mg-IV
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 6
mL/day | 139 (NA) — Standard deviation was not calculated due to limited sample size (n=2). Two out of five participants received only one dose and 1 participant had insufficient data. | 351 (177) | 181 (44.5) | 457 (214) | 180 (41.5)

11. Secondary Outcome: Terminal Elimination Half-life (t1/2) of MEDI-551
Description: The terminal elimination half-life (t1/2) was estimated based on the plasma concentrations of MEDI-551.
Time Frame: as for outcome 5
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | MEDI-551 30 Mg-IV | MEDI-551 60 Mg-SC | MEDI-551 100 Mg-IV | MEDI-551 300 Mg-SC | MEDI-551 600 Mg-IV
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 6
Day | 17.7 (NA) — Standard deviation was not calculated due to limited sample size (n=2). Two out of five participants received only one dose and 1 participant had insufficient data. | 12.3 (1.71) | 17.7 (6.27) | 15.1 (4.31) | 18.7 (2.03)

12. Secondary Outcome: Absolute Subcutaneous Bioavailability (F%) of MEDI-551
Description: Bioavailability (F%) is the fraction of the study drug absorbed through non-intravenous administration compared with the corresponding intravenous administration of the same drug.
Time Frame: Predose (Day 1) and Days 4, 8, 15, 29, 57, 85, 113, 141, and 169
Population: Safety Population
Measure: Number; unit: Percentage of bioavailability
Arm/Group | MEDI-551 60 Mg-SC | MEDI-551 300 Mg-SC
Number analyzed (Participants) | 3 | 3
Percentage of bioavailability | 58 | 46

13. Secondary Outcome: Absolute CD20 B-cell Count at Baseline
Description: Baseline absolute CD20 count is measured as the average between screening and predose on Day 1.
Time Frame: Baseline (Days -28 to -1)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: cells/mcL
Arm/Group | PLACEBO-IV-SC | MEDI-551 30 Mg-IV | MEDI-551 60 Mg-SC | MEDI-551 100 Mg-IV | MEDI-551 300 Mg-SC | MEDI-551 600 Mg-IV
Number analyzed (Participants) | 7 | 5 | 3 | 4 | 3 | 6
cells/mcL | 190 (99.1) | 173 (36.1) | 180 (108) | 183 (65.5) | 366 (257) | 201 (91.3)

14. Secondary Outcome: Time to 90 Percent (%) CD20 B-cell Depletion
Description: Time in days of first observation where CD20 counts fall to or below 10 percent (%) of baseline.
Time Frame: Baseline (Days -28 to -1) to long-term follow-up (LTFU) (Up to 18 months after EDV or 24 Week treatment period)
Population: Safety Population. No participants in placebo-IV-SC group reached 90% CD20 B-cell depletion.
Measure: Median (Full Range); unit: Day
Arm/Group | PLACEBO-IV-SC | MEDI-551 30 Mg-IV | MEDI-551 60 Mg-SC | MEDI-551 100 Mg-IV | MEDI-551 300 Mg-SC | MEDI-551 600 Mg-IV
Number analyzed (Participants) | 0 | 5 | 3 | 4 | 3 | 6
Day |  | 15.0 (1.10) [13.0 to 16.0] | 88.0 (50.3) [4.00 to 94.0] | 25.0 (6.19) [15.0 to 29.0] | 15.0 (4.04) [15.0 to 22.0] | 14.5 (5.65) [4.00 to 17.0]

15. Secondary Outcome: Duration of Suppression Greater Than or Equal to 90 % of CD20 B-cell Count
Description: Time in days of last observation where CD20 counts remain at or below 10% of baseline. Participants whose samples are available were analyzed for this outcome measure.
Time Frame: Baseline (Days -28 to -1) to LTFU (Up to 18 months after EDV or 24 Week treatment period)
Population: Safety Population. No participants were included in placebo-IV-SC group since no participant reached 90% depletion.
Measure: Median (Full Range); unit: Day
Arm/Group | PLACEBO-IV-SC | MEDI-551 30 Mg-IV | MEDI-551 60 Mg-SC | MEDI-551 100 Mg-IV | MEDI-551 300 Mg-SC | MEDI-551 600 Mg-IV
Number analyzed (Participants) | 0 | 4 | 2 | 4 | 3 | 5
Day |  | 149 (62.8) [69.0 to 200] | 100 (28.3) [77.0 to 123] | 180 (39.2) [140 to 229] | 211 (17.3) [175 to 213] | 254 (45.3) [244 to 332]

16. Secondary Outcome: Maximum Change From Baseline in Absolute CD20 of Peripheral Blood B-cell Count to LTFU
Description: The maximum degree of depletion (intensity) measured during the course of the study for each participant by subtracting 100 from the lowest observed percent of baseline value.
Time Frame: Baseline (Days -28 to -1) to LTFU (Up to 18 months after EDV or 24 Week treatment period)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percentage of cells
Arm/Group | PLACEBO-IV-SC | MEDI-551 30 Mg-IV | MEDI-551 60 Mg-SC | MEDI-551 100 Mg-IV | MEDI-551 300 Mg-SC | MEDI-551 600 Mg-IV
Number analyzed (Participants) | 7 | 5 | 3 | 4 | 3 | 6
Percentage of cells | 25.0 (31.2) | 99.8 (0.0770) | 99.2 (0.787) | 99.7 (0.225) | 99.8 (0.182) | 99.8 (0.237)

17. Secondary Outcome: Number of Participants Positive for Anti-Drug Antibodies to MEDI-551
Description: A participant was considered anti-drug antibody positive across the study if they had a positive reading at any time point during the study.
Time Frame: Days 1, 29, 85 and 169
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | PLACEBO-IV-SC | MEDI-551 30 Mg-IV | MEDI-551 60 Mg-SC | MEDI-551 100 Mg-IV | MEDI-551 300 Mg-SC | MEDI-551 600 Mg-IV
Number analyzed (Participants) | 7 | 5 | 3 | 4 | 3 | 6
Participants
  Day 1 (Baseline) | 0 | 0 | 0 | 0 | 0 | 0
  Day 29 | 0 | 0 | 0 | 0 | 0 | 0
  Day 85 | 0 | 0 | 0 | 0 | 0 | 0
  Day 169 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs were collected from the time of signature on informed consent through Day 169, SAEs were collected upto the long-term follow-up period (up to 18 months after early discontinuation visit or 24-week treatment period).
Arm/Group | PLACEBO-IV-SC | MEDI-551 60 Mg-SC | MEDI-551 100 Mg-IV | MEDI-551 300 Mg-SC | MEDI-551 30 Mg-IV | MEDI-551 600 Mg-IV
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/3 | 0/4 | 1/3 | 1/5 | 1/6
Other Adverse Events (participants affected / at risk) | 5/7 | 3/3 | 3/4 | 2/3 | 4/5 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO-IV-SC (N=7) | MEDI-551 60 Mg-SC (N=3) | MEDI-551 100 Mg-IV (N=4) | MEDI-551 300 Mg-SC (N=3) | MEDI-551 30 Mg-IV (N=5) | MEDI-551 600 Mg-IV (N=6)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Multiple sclerosis relapse (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO-IV-SC (N=7) | MEDI-551 60 Mg-SC (N=3) | MEDI-551 100 Mg-IV (N=4) | MEDI-551 300 Mg-SC (N=3) | MEDI-551 30 Mg-IV (N=5) | MEDI-551 600 Mg-IV (N=6)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (8) | 0 (0) | 1 (3) | 0 (0) | 2 (3) | 3 (6)
Blood pressure increased (Investigations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Multiple sclerosis relapse (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract inflammation (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.